CLINICAL TRIAL: NCT01570725
Title: A Portable Virtual Reality System as an Alternative Medical Treatment to Reduce Anxiety in Ambulatory Surgical Operations: a Randomized Controlled Study
Brief Title: Virtual Reality to Reduce Anxiety in Ambulatory Surgical Operations
Acronym: VRSurg
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting the selected subjects
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: VR01
Record Dates: First submitted 2009-02-22; First posted 2012-04-04 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Anxiety
Keywords: Immersive virtual reality; e-health; surgery; anxiety; relaxation; Patients who undergo ambulatory surgical operations
MeSH Terms: conditions — Anxiety Disorders | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Virtual reality exposure to a relaxing virtual environment. The virtual experience will be provided using immersive equipment.
  Interventions: Behavioral: Virtual reality exposure
- 2 (Experimental): Exposure to relaxing music. The music will be selected between classical music tunes.
  Interventions: Behavioral: Music only

INTERVENTIONS:
Behavioral: Virtual reality exposure — The Green Valley, a non interactive, relaxing environment showing a mountain landscape around a calm lake is presented to the patient together with the relaxing music and soft sounds (birds' songs, the water flowing, etc). Having the impression of walking around the lake, patients can observe the nature and virtually seat on a comfortable deck chair, in order to become easily relaxed.
  Patients were exposed to the virtual environment for the entire length of the operation.
  Arms: 1
Behavioral: Music only — A relaxing music and nature sounds have been used to provide a calm atmosphere and reduce stress. In the Music group it was provided to the patients through earphones with no visual stimulation.
  Arms: 2

SUMMARY:
Background. Preoperative anxiety is a common problem for patients who undergo surgical operations, being often associated with a number of negative behaviours during and after the surgical experience. Since drug treatments alone have frequently proved to be inadequate to reduce stress and anxiety in surgical contexts, in the last decades there has been an increased interest in non invasive complementary and alternative medical therapies (CAM), including music, relaxation, guided imagery, hypnosis, etc. that reduce pain and tension during pre and post operative phases. Virtual reality can be considered an innovative form of e-health-based CAM therapy having gained recognition as a means of attenuating pain during medical procedures. VR reduces distress and pain perception by providing a particularly intense form of immersive distraction that taxes the patient's limited attention capacity, resulting in the withdrawal of attention from the real, noxious, external stimulus with a subsequent reduction in pain and stress.

Objective. The aim of this study is to test the efficacy of a small, portable and immersive virtual reality system to reduce anxiety in a sample of patients who underwent ambulatory surgical operations under local or regional anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* all patients who undergo ambulatory surgical operations and sign informed consent

Exclusion Criteria:

* death or blind patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Psychological measure of anxiety (VAS-A) | One day before operation; one hour after operation; one week after operation
  Change from baseline in the level of anxiety

SECONDARY OUTCOMES:
Physiological parameter (heart rate) | One day before operation; one hour after operation; one week after operation
  Change from baseline in the heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Riva, PHD, Study Director — Istituto Auxologico Italiano
Locations (1):
- Regional Hospital No. 25 of the IMSS, Mexico City, Mexico